CLINICAL TRIAL: NCT01639001
Title: PHASE 3, RANDOMIZED, OPEN-LABEL STUDY OF THE EFFICACY AND SAFETY OF CRIZOTINIB VERSUS PEMETREXED/CISPLATIN OR PEMETREXED/CARBOPLATIN IN PREVIOUSLY UNTREATED EAST ASIAN PATIENTS WITH NON-SQUAMOUS CARCINOMA OF THE LUNG HARBORING A TRANSLOCATION OR INVERSION EVENT INVOLVING THE ANAPLASTIC LYMPHOMA KINASE (ALK) GENE LOCUS
Brief Title: A Study Of Crizotinib Versus Chemotherapy In Previously Untreated ALK Positive East Asian Non-Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8081029
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
Keywords: Crizotinib; ALK positive; ALK; Anaplastic Lymphoma Kinase; NSCLC; Non-Small Cell Lung Cancer; Frontline; 1L; Previously Untreated; East Asian; Non-Squamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crizotinib (Experimental): Crizotinib
  Interventions: Drug: Crizotinib
- Chemotherapy (Active Comparator): Chemotherapy [Option at Investigator's Choice]
  Interventions: Drug: Pemetrexed/Cisplatin; Drug: Pemetrexed/Carboplatin

INTERVENTIONS:
Drug: Crizotinib — 250 mg two times daily [BID], oral, on a continuous daily dosing schedule. Cycles are defined in 21 day periods.
  Arms: Crizotinib
Drug: Pemetrexed/Cisplatin — Option 1: Pemetrexed/Cisplatin; Pemetrexed, 500 mg/m^2, will be administered by intravenous infusion over 10 minutes or according to institutional administration timing on Day 1 of a 21-day cycle. Cisplatin, 75 mg/m^2 will be administered by infusion after adequate hydration according to institutional practices beginning approximately 30 minutes after the end of the pemetrexed infusion. Pemetrexed and cisplatin will be repeated every 3 weeks for a maximum of 6 cycles.
  Arms: Chemotherapy
Drug: Pemetrexed/Carboplatin — Option 2: Pemetrexed/Carboplatin. Pemetrexed, 500 mg/m^2, will be administered by intravenous infusion over 10 minutes or according to institutional administration timing on Day 1 of a 21-day cycle. Carboplatin, at a dose calculated to produce an AUC of 5 or 6 mg.min/mL will be administered by infusion according to institutional practices beginning approximately 30 minutes after the end of the pemetrexed infusion. Pemetrexed and carboplatin will be repeated every 3 weeks for a maximum of 6 cycles.
  Arms: Chemotherapy

SUMMARY:
This is a Phase III, Randomized, Open-label, Efficacy and Safety Study of Crizotinib single agent versus Chemotherapy Regimens (Pemetrexed/Cisplatin or Pemetrexed/Carboplatin) in First-Line ALK (Anaplastic Lymphoma Kinase) Positive East Asian Non-Small Cell Lung Cancer Patients. The objective of the study is to demonstrate that Crizotinib is superior to first-line chemotherapy pemetrexed/cisplatin or pemetrexed/carboplatin in prolonging Progression Free Survival (PFS) in East Asian patients with advanced Non-Squamous NSCLC whose tumors harbor a translocation or inversion event involving the ALK (Anaplastic Lymphoma Kinase) gene locus.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of locally advanced not suitable for local treatment, recurrent and metastatic non-squamous cell carcinoma of the lung.
* Positive for translocation or inversion events involving the ALK gene locus.
* No prior systemic treatment for locally advanced or metastatic disease. Patients with brain metastases only if treated and neurologically stable for at least 2 weeks and are not taking any medications contraindicated in Exclusion Criteria
* Evidence of a personally signed and dated informed consent document and willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures including completion of patient reported outcome [PRO] measures.

Exclusion Criteria:

* Current treatment on another therapeutic clinical trial.
* Prior therapy directly targeting ALK.
* Any of the following within the 3 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack. Appropriate treatment with anticoagulants is permitted.
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade >=2, uncontrolled atrial fibrillation of any grade, or QTc interval >470 msec.
* Pregnancy or breastfeeding.
* Use of drugs or foods that are known potent CYP3A inducers/inhibitors Concurrent use of drugs that are CYP3A substrates with narrow therapeutic indices.
* Known HIV infection
* History of extensive disseminated/bilateral or known presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis, but not history of prior radiation pneumonitis.
* Other severe acute or chronic medical conditions (including severe gastrointestinal conditions such as diarrhea or ulcer) or psychiatric conditions, or end-stage renal disease on hemodialysis, or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, and which would, therefore, make the patient inappropriate for entry into this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2012-09-29 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- China (34):
  - The First Affiliated Hospital of Anhui Medical University, Department of Medical Oncology, Hefei, Anhui
  - Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Dept. of Respiration. Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Oncology Department, the Second Affiliated Hospital of Third Military Medical University,PLA, Chongqing, Chongqing Municipality
  - Oncology Department, XinQiao Hospital of Third Military Medical University,, Chongqing, Chongqing Municipality
  - Fujian Province Oncology Hospital, Fuzhou, Fujian
  - SUN Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong General Hospital, Oncology Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical College/Thoracic Surgery, Guangzhou, Guangdong
  - Department 2 of Chemotherapy, Tumour Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology/Cancer Center, Wuhan, Hubei
  - Hunan Provincial Tumor Hospital/Division of Oncology, Changsha, Hunan
  - Nanjing General Hospital of Nanjing Military Command, Department of Respiratory medicine, Nanjing, Jiangsu
  - Department of Oncology, Jilin Provincial Cancer Hospital, Changchun, Jilin
  - The first hospital of China Medical University/Oncology Department, Shenyang, Liaoning
  - Oncology Department, West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Province Cancer Hospital/Department of Pulmonary Tumor, Chengdu, Sichuan
  - Department of Respiratory, The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of College of Medicine of Zhejiang University, Center for Oncology, Hangzhou, Zhejiang
  - 307 Hospital of PLA/Department of Lung Cancer, Beijing
  - Beijing Cancer Hospital, Beijing
  - The Military General Hospital of Beijing PLA, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Respiration department,the First Affiliated Hospital of Third Military Medical University, PLA, Chongqing
  - Shanghai Chest Hospital/Lung cancer clinical center, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University / Respiratory Department, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Malaysia (2):
  - Department of Nuclear Medicine, Radiotherapy and Oncology, Hospital Universiti Sains Malaysia, Kubang Kerian, Kota Bahru, Kelantan
  - Hospital Pulau Pinang, George Town, Pulau Pinang
- Taiwan (5):
  - Chi Mei Medical Center Liouying, Liou Ying Township, Tainan
  - Chung Shan Medical University Hospital, Taichung
  - Chi Mei Medical Center Liuying, Tainan
  - Taipei Veterans General Hospital, Chest Department, Taipei
  - Chang Gung Medical Foundation, LinKou Branch, Taoyuan District
- Thailand (2):
  - Medical Oncology Unit, Department of Medicine, Faculty of Medicine, Chulalongkorn University, Pathumwan, Bangkok
  - Division of Medical Oncology, Department of Medicine, Faculty of Medicine, Siriraj Hospital,, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wu YL, Lu S, Lu Y, Zhou J, Shi YK, Sriuranpong V, Ho JCM, Ong CK, Tsai CM, Chung CH, Wilner KD, Tang Y, Masters ET, Selaru P, Mok TS. Results of PROFILE 1029, a Phase III Comparison of First-Line Crizotinib versus Chemotherapy in East Asian Patients with ALK-Positive Advanced Non-Small Cell Lung Cancer. J Thorac Oncol. 2018 Oct;13(10):1539-1548. doi: 10.1016/j.jtho.2018.06.012. Epub 2018 Aug 14. PMID 29966800
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081029&StudyName=A%20Study%20Of%20Crizotinib%20Versus%20Chemotherapy%20In%20Previously%20Untreated%20ALK%20Positive%20East%20Asian%20Non-Small%20Cell%20Lung%20Cancer%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 3, randomized, open label, multicenter study conducted in 35 centers in 5 countries. A total of 207 actual participants were randomized, 104 in the crizotinib arm and 103 in the chemotherapy (pemetrexed/cisplatin or pemetrexed/carboplatin) arm.
Pre-assignment Details: Participants with histologically or cytologically proven diagnosis of locally advanced, recurrent, or metastatic non squamous non small cell lung cancer and tumors with measurable disease were enrolled. Participants were to be positive for translocation or inversion events involving the ALK gene locus as determined by an ALK break-apart FISH test.
Groups:
- Crizotinib: Crizotinib capsules, 250 mg twice daily (BID), were administered orally at approximately the same time each day on a continuous daily dosing schedule. Each treatment cycle was defined as 21 days. Participants could continue crizotinib treatment beyond the time of RECIST defined Progressive Disease (PD), as determined by independent radiology review (IRR), at the discretion of the investigator if the participant was perceived to be experiencing clinical benefit. The maximum duration of crizotinib treatment was 324.4 weeks.
- Chemotherapy: Standard doses of chemotherapy were administered by intravenous (IV) infusion every 3 weeks for a maximum of 6 cycles. Pemetrexed (500 mg/m2) was administered over 10 minutes or according to institutional administration timing; cisplatin (75 mg/m2) was administered after adequate hydration beginning approximately 30 minutes after the end of the pemetrexed infusion and carboplatin was administered on Day 1 of a 21-day cycle at a dose calculated to produce an area under the concentration time curve [AUC] of 5 or 6 mg*min/mL, beginning approximately 30 minutes after end of pemetrexed infusion. The maximum duration of chemotherapy treatment was 24.1 weeks.
Period: Overall Study
Arm/Group | Crizotinib | Chemotherapy
Started | 104 | 103
Treated | 104 | 101
Completed ("Completed" refers to either those patients who switched to commercial supplies of crizotinib or those patients who were in survival follow up, when the Sponsor sent a written End of Study notification to the study sites.) | 29 | 26
Not Completed | 75 | 77
Not completed — Refused further follow-up | 9 | 12
Not completed — Lost to Follow-up | 3 | 0
Not completed — Death | 62 | 61
Not completed — Randomized but not treated | 0 | 2
Not completed — Long-term follow-up participants who did not respond to the contact from their study sites. | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crizotinib | Chemotherapy | Total
Number analyzed (Participants) | 104 | 103 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (10.6) | 48.9 (11.2) | 48.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 60 | 114
  Male | 50 | 43 | 93

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Based on IRR by Treatment Arm
Description: PFS was defined as the time from the date of randomization to the date of the first documentation of objective tumor progression (by IRR) or death on study due to any cause, whichever occured first. If tumor progression data included more than 1 date, the first date was used. PFS (in months) was calculated as (first event date - randomization date +1)/30.44. Progression is defined using RECIST v1.1, as at least a 20% increase (including an absolute increase of at least 5 millimeters) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: Randomization to objective progression, death or last tumor assessment without progression before any additional anti-cancer therapy (whichever occurred first, assessed up to 33 months)
Population: The Full Analysis (FA) population included all participants who were randomized with study treatment assignment designated according to the initial randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 103
Months | 11.1 [8.3 to 12.6] | 6.8 [5.7 to 7.0]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; The study was designed to test the null hypothesis H0: λ=1.0 versus the alternative hypothesis HA: λ < 1.0, where λ is the hazard ratio (HR; Crizotinib/Chemotherapy). Evaluation of 160 PFS events in the 2 arms using a 1-sided log-rank test at the 0.025 level of significance was required to detect a HR of 0.64 with 80% power; Test type: Superiority or Other; p < 0.0001, 1 sided stratified log-rank — The study was to be considered positive if the 1-sided log-rank test for PFS, stratified for baseline stratification factors (ECOG PS, ethnicity, and brain metastases) was significant at the 0.02496level; Hazard Ratio (HR) = 0.402, 95% CI 2-sided [0.286 to 0.565] — Based on the Cox Proportional hazards model stratified by ECOG PS, ethnicity, and brain metastases. Assuming proportional hazards, a hazard ratio less than 1 indicates a reduction in hazard rate in favor of crizotinib

2. Secondary Outcome: Objective Response Rate (ORR) - Percentage of Participants With Objective Response Based on IRR
Description: Percentage of participants with objective response of complete response (CR) or partial response (PR) according to RECIST version 1.1. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Randomization to objective progression, death or last tumor assessment without progression before any additional anti-cancer therapy (assessed up to 33 months)
Population: FA population included all participants who were randomized with study treatment assignment designated according to the initial randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 103
Percentage of participants | 87.5 [79.6 to 93.2] | 45.6 [35.8 to 55.7]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; The confidence interval for the treatment difference was based on normal distribution; Test type: Superiority or Other; p < 0.0001, 2-sided pearson chi-square test — If the PFS endpoint was significant, ORR was to be considered significant if 2-sided p-value from Pearson chi-square test was <= 0.04992; Treatment Difference = 41.869, 95% CI 2-sided [30.340 to 53.398] — Treatment difference in ORR (%)

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death due to any cause. OS (in months) was calculated as (date of death - date of randomization +1)/30.44. For participants who were lost to follow-up or withdrew consent, the OS was censored on the last date that participants were known to be alive.
Time Frame: From randomization to death or last date known as alive for those who were lost to follow-up or withdrew consent (assessed up to 64 months).
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 103
Months | 33.7 [26.5 to 42.5] | 32.9 [23.9 to 43.1]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Test type: Superiority or Other; p = 0.6172, 1 sided stratified log-rank — If the PFS and ORR endpoints were significant, OS was to be considered significant if 1-sided, log-rank test stratified for ECOG, ethnicity and metastases was <= 0.02496; Hazard Ratio (HR) = 1.056, 95% CI 2-sided [0.734 to 1.521] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With Disease Control at 12 Weeks Based on IRR
Description: Disease Control Rate (DCR) at 12 weeks is defined as the percent of participants with CR, PR or stable disease (SD) at 12 weeks according to RECIST version 1.1 as determined by the IRR. The best response of SD can be assigned if SD criteria were met at least once after randomization at a minimum interval of 6 weeks. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions and disappearance of all non-target lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: From randomization to Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 103
Percentage of participants | 82.7 [74.0 to 89.4] | 73.8 [64.2 to 82.0]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; The confidence interval for the treatment difference was based on normal distribution; Test type: Superiority or Other; p = 0.1204, 2-sided pearson chi-square test; Treatment difference = 8.906, 95% CI 2-sided [-2.275 to 20.086] — Treatment Difference in DCR Rate (%)

5. Secondary Outcome: Estimate of the Percentage of Participants Surviving at 1 Year and at 18 Months
Description: Probability of survival 1 year and 18 month after randomization. The probability of survival at 1 year was estimated using the Kaplan Meier method and a 2-sided 95% CI for the log [-log(1-year survival probability)] was calculated using a normal approximation and then back transformed to give a CI for the 1-year survival probability itself. The probability of survival at 18 months was estimated similarly.
Time Frame: From randomization to 1 year and from randomization to 18 months
Population: The FA population included all participants who were randomized with study treatment assignment designated according to the initial randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of paricipants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 103
Percentage of paricipants
  Up to 1 year | 79.3 [70.0 to 86.0] | 79.5 [70.0 to 86.3]
  Up to 18 months | 71.2 [61.2 to 79.0] | 72.1 [62.0 to 79.9]

6. Secondary Outcome: Duration of Response (DR) Based on IRR
Description: DR was defined as the time from the first documentation of objective tumor response (CR or PR), as determined by the IRR, to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. DR (in weeks) was calculated as (first date of PD or death - first date of CR or PR +1)/7. DR was only calculated for the subgroup of participants with an objective tumor response.
Time Frame: From objective response to date of progression, death or last tumor assessment without progression before any additional anti-cancer therapy (whichever occurred first, up to 33 months)
Population: FA population included all participants who were randomized with study treatment assignment designated according to the initial randomization. N = Participants with objective tumor response by IRR.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 91 | 47
Weeks | 44.4 [35.9 to 60.0] | 18.1 [16.7 to 19.9]

7. Secondary Outcome: Time to Tumor Response (TTR) Based on IRR
Description: TTR was defined as the time from randomization to first documentation of objective tumor response (CR or PR) as determined by the IRR. For participants proceeding from PR to CR, the onset of PR was taken as the onset of response. TTR was calculated for the subgroup of participants with objective tumor response.
Time Frame: Randomization to first documentation of objective tumor response (up to 33 months).
Population: FA population included all participants who were randomized with study treatment assignment designated according to the initial randomization. N=Participants who had objective tumor response by IRR.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 91 | 47
Weeks | 6.3 [5.1 to 24.9] | 12.1 [5.7 to 36.1]

8. Secondary Outcome: Time to Progression (TTP) Based on IRR
Description: TTP was defined as the time from the date of randomization to the date of the first documentation of objective tumor progression, as determined by IRR. If tumor progression data included more than 1 date, the first date was used. TTP (in months) was calculated as (first event date - randomization date +1)/30.44.
Time Frame: Randomization to objective progression, death or last tumor assessment without progression before any additional anti-cancer therapy (whichever occurred first, up to 33 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 103
Months | 12.0 [8.4 to 15.4] | 6.9 [5.7 to 7.1]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Test type: Superiority or Other; p < 0.0001, 1 sided unstratified log-rank; Hazard Ratio (HR) = 0.348, 95% CI 2-sided [0.246 to 0.493] — Based on the Cox Proportional hazards model

9. Secondary Outcome: Intracranial Time to Progression (IC-TTP) Based on IRR
Description: IC-TTP was defined similarly to TTP, but only considering intracranial disease (excluding extracranial disease) and the progression was determined based on either new brain metastases or progression of existing brain metastases.
Time Frame: Randomization to objective intracranial progression or last tumor assessment without progression before any additional anti-cancer therapy (whichever occurred first, up to 33 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 103
Months | NA [20.8 to NA] — Median and upper limit for IC-TTP was not reached due to insufficient IC-TTP events. | 16.0 [12.6 to NA] — Upper limit for IC-TTP was not reached due to insufficient IC-TTP events.
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Test type: Superiority or Other; p = 0.1270, 1 sided unstratified log-rank; Hazard Ratio (HR) = 0.669, 95% CI 2-sided [0.335 to 1.338] — Based on the Cox Proportional hazards model

10. Secondary Outcome: Extracranial Time to Progression (EC-TTP) Based on IRR
Description: EC-TTP was defined similarly to TTP, but only considering extracranial disease (excluding intracranial disease) and the progression was determined based on either new extracranial lesions or progression of existing extracranial lesions.
Time Frame: Randomization to objective extracranial progression or last tumor assessment without progression before any additional anti-cancer therapy (whichever occurred first, up to 33 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 103
Months | 18.0 [12.3 to 20.9] | 7.0 [6.0 to 7.1]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Test type: Superiority or Other; p < 0.0001, 1 sided unstratified log-rank; Hazard Ratio (HR) = 0.277, 95% CI 2-sided [0.186 to 0.412] — Based on the Cox Proportional hazards model

11. Secondary Outcome: Time to Deterioration (TTD) in Participant Reported Pain, Dyspnea, or Cough Assessed Using Quality of Life Questionnaire Supplement Module for Lung Cancer (QLQ-LC13)
Description: The QLQ-LC13 consisted of 1 multi-item scale and 9 single items that assessed the specific symptoms (dyspnea, cough, hemoptysis, and site specific pain), side effects (sore mouth, dysphagia, neuropathy, and alopecia), and pain medication use of lung cancer participants receiving chemotherapy. The QLQ-LC13 Coughing, Dyspnoea and Pain in chest each ranged from 0-100 with higher scores indicating a high level of symptomatology/problems. TTD in pain in chest, dyspnea, or cough from the QLQ-LC13 was a composite endpoint defined as the time from randomization to the earliest time the participant's scale scores showed a 10 point or greater increase after baseline in any of the 3 symptoms.
Time Frame: From Baseline to deterioration while on study treatment. For participants with no deterioration, the data was censored at the last date when QLQ-LC13 assessment for pain, dyspnea, or cough was completed (assessed up to 33 months）
Population: Participants from the safety analysis population who completed a baseline and at least 1 post-baseline PRO assessment for pain in chest, dyspnea or cough.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 103 | 98
Months | 2.8 [1.4 to 6.9] | 0.3 [0.3 to 0.5]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Test type: Superiority or Other; p < 0.0001, 2 sided unstratified log rank — 2-sided Hochberg adjusted p-values; Hazard Ratio (HR) = 0.432, 95% CI 2-sided [0.307 to 0.610] — Based on the Cox Proportional hazards model

12. Secondary Outcome: Change From Baseline in Functioning and Global Quality of Life (QOL) as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30)
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). The QLQ-C30 Global QOL, Physical Functioning, Role Functioning, Cognitive Functioning, Emotional Functioning, and Social Functioning each ranged from 0-100 with higher scores indicating a better level of functioning or better quality of life.
Time Frame: as for outcome 11
Population: Participants from the safety analysis population who completed a baseline and at least 1 post-baseline PRO assessment.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 103 | 98
Units on a scale
  QLQ-C30 Global QoL | 5.0891 [2.53 to 7.64] | -2.3619 [-5.00 to 0.28]
  QLQ-C30 Cognitive Functioning | -1.1896 [-3.28 to 0.90] | -4.8026 [-6.95 to -2.66]
  QLQ-C30 Emotional Functioning | 3.7077 [1.76 to 5.66] | 2.0557 [0.04 to 4.07]
  QLQ-C30 Physical Functioning | 3.7705 [1.97 to 5.57] | -2.9562 [-4.82 to -1.10]
  QLQ-C30 Role Functioning | 1.0538 [-1.56 to 3.66] | -5.7570 [-8.44 to -3.07]
  QLQ-C30 Social Functioning | 0.8712 [-2.27 to 4.02] | -4.7228 [-7.96 to -1.49]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 Global QoL. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 7.4510, 95% CI 2-sided [3.79 to 11.11]
Statistical Analysis 2: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 cognitive functioning. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0140, Mixed Models Analysis; Mean Difference (Net) = 3.6130, 95% CI 2-sided [0.73 to 6.49]
Statistical Analysis 3: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 emotional functioning. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.2427, Mixed Models Analysis; Mean Difference (Net) = 1.6520, 95% CI 2-sided [-1.12 to 4.42]
Statistical Analysis 4: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 physical functioning. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 6.7267, 95% CI 2-sided [4.15 to 9.30]
Statistical Analysis 5: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 role functioning. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Net) = 6.8109, 95% CI 2-sided [3.15 to 10.47]
Statistical Analysis 6: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 social functioning. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0140, Mixed Models Analysis; Mean Difference (Net) = 5.5940, 95% CI 2-sided [1.13 to 10.06]

13. Secondary Outcome: Change From Baseline Scores in QLQ-C30 Symptoms as Assessed by the EORTC-QLQ-C30
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). The QLQ-C30 Appetite loss, Constipation, Diarrhea, Dyspnea, Fatigue, Financial difficulties, Insomnia, Nausea/vomiting, and Pain each ranged from 0-100 with higher scores indicating a high level of symptomatology/problems.
Time Frame: as for outcome 11
Population: Participants from the safety analysis population who completed a baseline and at least 1 post-baseline PRO assessment.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 103 | 98
Units on a scale
  QLQ-C30 Appetite loss | -1.5967 [-4.18 to 0.99] | 4.4465 [1.74 to 7.15]
  QLQ-C30 Constipation | 7.1367 [4.40 to 9.87] | 2.6341 [-0.23 to 5.50]
  QLQ-C30 Diarrhea | 15.3294 [13.35 to 17.31] | -0.4791 [-2.55 to 1.60]
  QLQ-C30 Dyspnea | -7.9353 [-10.41 to -5.46] | -0.1903 [-2.75 to 2.37]
  QLQ-C30 Fatigue | -3.8888 [-6.20 to -1.58] | 2.6028 [0.21 to 5.00]
  QLQ-C30 Financial Difficulties | -3.2339 [-7.26 to 0.79] | 0.3826 [-3.74 to 4.51]
  QLQ-C30 Insomnia | -8.3816 [-10.95 to -5.81] | -1.6060 [-4.29 to 1.07]
  QLQ-C30 Nausea and Vomiting | 4.0796 [2.06 to 6.09] | 6.5986 [4.48 to 8.72]
  QLQ-C30 Pain | -9.1305 [-11.27 to -6.99] | -0.6956 [-2.90 to 1.51]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 appetite loss. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; Mean Difference (Net) = -6.0432, 95% CI 2-sided [-9.79 to -2.30]
Statistical Analysis 2: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 constipation. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0263, Mixed Models Analysis; Mean Difference (Net) = 4.5026, 95% CI 2-sided [0.53 to 8.47]
Statistical Analysis 3: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 diarrhea. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 15.8085, 95% CI 2-sided [12.94 to 18.68]
Statistical Analysis 4: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 dyspnea. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -7.7449, 95% CI 2-sided [-11.30 to -4.19]
Statistical Analysis 5: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 fatigue. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Net) = -6.4915, 95% CI 2-sided [-9.82 to -3.17]
Statistical Analysis 6: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 financial difficulties. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.2099, Mixed Models Analysis; Mean Difference (Net) = -3.6165, 95% CI 2-sided [-9.27 to 2.04]
Statistical Analysis 7: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 insomnia. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Net) = -6.7756, 95% CI 2-sided [-10.49 to -3.06]
Statistical Analysis 8: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 nausea and vomiting. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0902, Mixed Models Analysis; Mean Difference (Net) = -2.5190, 95% CI 2-sided [-5.43 to 0.40]
Statistical Analysis 9: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-C30 pain. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -8.4349, 95% CI 2-sided [-11.42 to -5.45]

14. Secondary Outcome: Change From Baseline in Lung Cancer Symptom Scores as Assessed by the EORTC Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13)
Description: The QLQ-LC13 consisted of 1 multi-item scale and 9 single items that assessed the specific symptoms (dyspnea, cough, hemoptysis, and site specific pain), side effects (sore mouth, dysphagia, neuropathy, and alopecia), and pain medication use of lung cancer participants receiving chemotherapy. The QLQ-LC13 Alopecia, Coughing, Dysphagia, Dyspnoea, Haemoptysis, Pain in arm or shoulder, Pain in chest, Pain in other parts, Peripheral neuropathy, and Sore mouth each ranged from 0-100 with higher scores indicating a high level of symptomatology/problems.
Time Frame: as for outcome 11
Population: Participants from the safety analysis population who completed a baseline and at least 1 post-baseline PRO assessment.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 103 | 98
Units on a scale
  QLQ-LC13 Alopecia | -2.0837 [-4.41 to 0.24] | 2.7710 [0.37 to 5.18]
  QLQ-LC13 Coughing | -17.2704 [-19.96 to -14.58] | -10.2748 [-13.07 to -7.48]
  QLQ-LC13 Dysphagia | 0.5354 [-1.34 to 2.41] | 1.0535 [-0.90 to 3.01]
  QLQ-LC13 Dyspnoea | -9.0842 [-11.34 to -6.83] | -0.4371 [-2.76 to 1.89]
  QLQ-LC13 Haemoptysis | -4.3017 [-5.42 to -3.18] | -3.0513 [-4.22 to -1.88]
  QLQ-LC13 Pain in Arm or Shoulder | -6.8289 [-9.43 to -4.23] | -2.5927 [-5.29 to 0.11]
  QLQ-LC13 Pain in Chest | -8.3565 [-10.81 to -5.90] | -4.1328 [-6.68 to -1.58]
  QLQ-LC13 Pain in Other Parts | -4.8475 [-7.22 to -2.48] | -0.2573 [-2.72 to 2.21]
  QLQ-LC13 Peripheral Neuropathy | 0.1787 [-1.94 to 2.30] | 1.8519 [-0.36 to 4.06]
  QLQ-LC13 Sore Mouth | 1.5134 [-0.01 to 3.03] | 3.9114 [2.30 to 5.53]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 alopecia. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0039, Mixed Models Analysis; Mean Difference (Net) = -4.8547, 95% CI 2-sided [-8.15 to -1.56]
Statistical Analysis 2: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 coughing. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Net) = -6.9957, 95% CI 2-sided [-10.85 to -3.14]
Statistical Analysis 3: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 dysphagia. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.7082, Mixed Models Analysis; Mean Difference (Net) = -0.5181, 95% CI 2-sided [-3.23 to 2.20]
Statistical Analysis 4: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 dyspnoea. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -8.6471, 95% CI 2-sided [-11.85 to -5.44]
Statistical Analysis 5: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 haemoptysis. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.1284, Mixed Models Analysis; Mean Difference (Net) = -1.2504, 95% CI 2-sided [-2.86 to 0.36]
Statistical Analysis 6: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 pain in arm or shoulder. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0265, Mixed Models Analysis; Mean Difference (Net) = -4.2363, 95% CI 2-sided [-7.98 to -0.49]
Statistical Analysis 7: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 pain in chest. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0185, Mixed Models Analysis; Mean Difference (Net) = -4.2237, 95% CI 2-sided [-7.74 to -0.71]
Statistical Analysis 8: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 pain in other parts. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0075, Mixed Models Analysis; Mean Difference (Net) = -4.5901, 95% CI 2-sided [-7.95 to -1.23]
Statistical Analysis 9: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 peripheral neuropathy. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.2848, Mixed Models Analysis; Mean Difference (Net) = -1.6732, 95% CI 2-sided [-4.74 to 1.39]
Statistical Analysis 10: Comparison: Crizotinib vs Chemotherapy; Analysis presented for QLQ-LC13 sore mouth. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EORTC QLQ-C30 subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0296, Mixed Models Analysis; Mean Difference (Net) = -2.3980, 95% CI 2-sided [-4.56 to -0.24]

15. Secondary Outcome: Change From Baseline in General Health Status as Assessed by EuroQol 5D (EQ-5D)-Visual Analog Scale (VAS)
Description: EQ-5D is a standardized, participant-administered measure of health outcome. It provides a descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), using 3 levels (no, moderate, or extreme problems) and a visual analog scale (VAS). The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: as for outcome 11
Population: Participants from the safety analysis population who completed a baseline and at least 1 post-baseline PRO assessment.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 102 | 98
Units on a scale | 3.4209 [1.20 to 5.64] | -0.4927 [-2.75 to 1.77]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; From a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EQ-5D VAS subscale score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0123, Mixed Models Analysis; Mean Difference (Net) = 3.9136, 95% CI 2-sided [0.85 to 6.98]

16. Secondary Outcome: Change From Baseline in General Health Status as Assessed by EQ-5D-Index
Description: EQ-5D is a standardized, participant-administered measure of health outcome. It provides a descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), using 3 levels (no, moderate, or extreme problems) and a visual analog scale (VAS). EQ-5D summary index is obtained with a formula that weights each level of the 5 dimensions. The index-based score is interpreted along a continuum of 0 (death) to 1 (perfect health).
Time Frame: From Baseline to deterioration while on study treatment. For participants with no deterioration, the data was censored at the last date when QLQ-LC13 assessment for pain, dyspnea, or cough was completed (assessed up to 33 months)
Population: Participants from the safety analysis population who completed a baseline and at least 1 post-baseline PRO assessment.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 102 | 98
Units on a scale | 0.0502 [0.02 to 0.08] | 0.0077 [-0.02 to 0.04]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; From a repeated measures mixed-effects model with an intercept term, treatment, visit day and baseline EQ-5D Index score (intercept and visit day are included as random effects). P-values and confidence intervals are not adjusted for multiplicity; Test type: Superiority or Other; p = 0.0320, Mixed Models Analysis; Mean Difference (Net) = 0.0425, 95% CI 2-sided [0.00 to 0.08]

17. Secondary Outcome: Percentage of Participants With Visual Disturbance as Assessed by Visual Symptom Assessment Questionnaire (VSAQ-ALK)
Description: VSAQ-ALK is a self-report measure that was developed to assess the problems of visual disturbances and symptoms may include the appearance of overlapping shadows and after images; shimmering, flashing or trailing lights; strings, streamers, or floaters; as well as hazy or blurry vision. The participants answered "Yes" to the first question (Q1) of VSAQ-ALK "Have you experienced any visual disturbances?" were considered to have experienced visual disturbance and were instructed to complete the rest of the questionnaire. The percentage of participants who responded to Q1 of VSAQ-ALK as "Yes" and as "No" during each study cycle was calculated as (n/N*)*100 where N* was the number of participants who had completed Q1.
Time Frame: Cycle 1 Day 1 to end of treatment or withdrawal, no later than 4 weeks (+/- 1 week) from last dose of study medication or when the decision was taken to withdraw from the study (whichever was sooner, assessed up to Cycle 86)
Population: Participants from the safety analysis population who completed a baseline and at least 1 post-baseline PRO assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 103 | 98
Percentage of participants
  Baseline: Cycle 1/Day 1 (Answer to Q1: Yes) | 6.8 | 7.1
  Baseline: Cycle 1/Day 1 (Answer to Q1: No) | 93.2 | 92.9
  Cycle 2/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 102 | 97
  Cycle 2/Day 1 (Answer to Q1: Yes) | 51.0 | 13.4
  Cycle 2/Day 1 (Answer to Q1: No): number analyzed (Participants) | 102 | 97
  Cycle 2/Day 1 (Answer to Q1: No) | 49.0 | 86.6
  Cycle 3/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 102 | 90
  Cycle 3/Day 1 (Answer to Q1: Yes) | 46.1 | 11.1
  Cycle 3/Day 1 (Answer to Q1: No): number analyzed (Participants) | 102 | 90
  Cycle 3/Day 1 (Answer to Q1: No) | 53.9 | 88.9
  Cycle 4/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 98 | 88
  Cycle 4/Day 1 (Answer to Q1: Yes) | 43.9 | 14.8
  Cycle 4/Day 1 (Answer to Q1: No): number analyzed (Participants) | 98 | 88
  Cycle 4/Day 1 (Answer to Q1: No) | 56.1 | 85.2
  Cycle 5/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 95 | 74
  Cycle 5/Day 1 (Answer to Q1: Yes) | 35.8 | 13.5
  Cycle 5/Day 1 (Answer to Q1: No): number analyzed (Participants) | 95 | 74
  Cycle 5/Day 1 (Answer to Q1: No) | 64.2 | 86.5
  Cycle 6/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 91 | 69
  Cycle 6/Day 1 (Answer to Q1: Yes) | 37.4 | 10.1
  Cycle 6/Day 1 (Answer to Q1: No): number analyzed (Participants) | 91 | 69
  Cycle 6/Day 1 (Answer to Q1: No) | 62.6 | 89.9
  Cycle 7/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 89 | 0
  Cycle 7/Day 1 (Answer to Q1: Yes) | 36.0 |
  Cycle 7/Day 1 (Answer to Q1: No): number analyzed (Participants) | 89 | 0
  Cycle 7/Day 1 (Answer to Q1: No) | 64.0 |
  Cycle 8/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 89 | 0
  Cycle 8/Day 1 (Answer to Q1: Yes) | 28.1 |
  Cycle 8/Day 1 (Answer to Q1: No): number analyzed (Participants) | 89 | 0
  Cycle 8/Day 1 (Answer to Q1: No) | 71.9 |
  Cycle 9/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 87 | 0
  Cycle 9/Day 1 (Answer to Q1: Yes) | 24.1 |
  Cycle 9/Day 1 (Answer to Q1: No): number analyzed (Participants) | 87 | 0
  Cycle 9/Day 1 (Answer to Q1: No) | 75.9 |
  Cycle 10/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 88 | 0
  Cycle 10/Day 1 (Answer to Q1: Yes) | 23.9 |
  Cycle 10/Day 1 (Answer to Q1: No): number analyzed (Participants) | 88 | 0
  Cycle 10/Day 1 (Answer to Q1: No) | 76.1 |
  Cycle 11/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 81 | 0
  Cycle 11/Day 1 (Answer to Q1: Yes) | 23.5 |
  Cycle 11/Day 1 (Answer to Q1: No): number analyzed (Participants) | 81 | 0
  Cycle 11/Day 1 (Answer to Q1: No) | 76.5 |
  Cycle 12/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 80 | 0
  Cycle 12/Day 1 (Answer to Q1: Yes) | 21.3 |
  Cycle 12/Day 1 (Answer to Q1: No): number analyzed (Participants) | 80 | 0
  Cycle 12/Day 1 (Answer to Q1: No) | 78.8 |
  Cycle 13/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 79 | 0
  Cycle 13/Day 1 (Answer to Q1: Yes) | 25.3 |
  Cycle 13/Day 1 (Answer to Q1: No): number analyzed (Participants) | 79 | 0
  Cycle 13/Day 1 (Answer to Q1: No) | 74.7 |
  Cycle 14/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 74 | 0
  Cycle 14/Day 1 (Answer to Q1: Yes) | 27.0 |
  Cycle 14/Day 1 (Answer to Q1: No): number analyzed (Participants) | 74 | 0
  Cycle 14/Day 1 (Answer to Q1: No) | 73.0 |
  Cycle 15/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 71 | 0
  Cycle 15/Day 1 (Answer to Q1: Yes) | 28.2 |
  Cycle 15/Day 1 (Answer to Q1: No): number analyzed (Participants) | 71 | 0
  Cycle 15/Day 1 (Answer to Q1: No) | 71.8 |
  Cycle 16/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 70 | 0
  Cycle 16/Day 1 (Answer to Q1: Yes) | 28.6 |
  Cycle 16/Day 1 (Answer to Q1: No): number analyzed (Participants) | 70 | 0
  Cycle 16/Day 1 (Answer to Q1: No) | 71.4 |
  Cycle 17/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 70 | 0
  Cycle 17/Day 1 (Answer to Q1: Yes) | 28.6 |
  Cycle 17/Day 1 (Answer to Q1: No): number analyzed (Participants) | 70 | 0
  Cycle 17/Day 1 (Answer to Q1: No) | 71.4 |
  Cycle 18/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 67 | 0
  Cycle 18/Day 1 (Answer to Q1: Yes) | 28.4 |
  Cycle 18/Day 1 (Answer to Q1: No): number analyzed (Participants) | 67 | 0
  Cycle 18/Day 1 (Answer to Q1: No) | 71.6 |
  Cycle 19/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 64 | 0
  Cycle 19/Day 1 (Answer to Q1: Yes) | 28.1 |
  Cycle 19/Day 1 (Answer to Q1: No): number analyzed (Participants) | 64 | 0
  Cycle 19/Day 1 (Answer to Q1: No) | 71.9 |
  Cycle 20/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 61 | 0
  Cycle 20/Day 1 (Answer to Q1: Yes) | 27.9 |
  Cycle 20/Day 1 (Answer to Q1: No): number analyzed (Participants) | 61 | 0
  Cycle 20/Day 1 (Answer to Q1: No) | 72.1 |
  Cycle 21/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 59 | 0
  Cycle 21/Day 1 (Answer to Q1: Yes) | 30.5 |
  Cycle 21/Day 1 (Answer to Q1: No): number analyzed (Participants) | 59 | 0
  Cycle 21/Day 1 (Answer to Q1: No) | 69.5 |
  Cycle 22/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 55 | 0
  Cycle 22/Day 1 (Answer to Q1: Yes) | 29.1 |
  Cycle 22/Day 1 (Answer to Q1: No): number analyzed (Participants) | 55 | 0
  Cycle 22/Day 1 (Answer to Q1: No) | 70.9 |
  Cycle 23/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 56 | 0
  Cycle 23/Day 1 (Answer to Q1: Yes) | 28.6 |
  Cycle 23/Day 1 (Answer to Q1: No): number analyzed (Participants) | 56 | 0
  Cycle 23/Day 1 (Answer to Q1: No) | 71.4 |
  Cycle 24/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 54 | 0
  Cycle 24/Day 1 (Answer to Q1: Yes) | 31.5 |
  Cycle 24/Day 1 (Answer to Q1: No): number analyzed (Participants) | 54 | 0
  Cycle 24/Day 1 (Answer to Q1: No) | 68.5 |
  Cycle 25/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 53 | 0
  Cycle 25/Day 1 (Answer to Q1: Yes) | 32.1 |
  Cycle 25/Day 1 (Answer to Q1: No): number analyzed (Participants) | 53 | 0
  Cycle 25/Day 1 (Answer to Q1: No) | 67.9 |
  Cycle 26/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 52 | 0
  Cycle 26/Day 1 (Answer to Q1: Yes) | 28.8 |
  Cycle 26/Day 1 (Answer to Q1: No): number analyzed (Participants) | 52 | 0
  Cycle 26/Day 1 (Answer to Q1: No) | 71.2 |
  Cycle 27/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 50 | 0
  Cycle 27/Day 1 (Answer to Q1: Yes) | 28.0 |
  Cycle 27/Day 1 (Answer to Q1: No): number analyzed (Participants) | 50 | 0
  Cycle 27/Day 1 (Answer to Q1: No) | 72.0 |
  Cycle 28/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 50 | 0
  Cycle 28/Day 1 (Answer to Q1: Yes) | 30.0 |
  Cycle 28/Day 1 (Answer to Q1: No): number analyzed (Participants) | 50 | 0
  Cycle 28/Day 1 (Answer to Q1: No) | 70.0 |
  Cycle 29/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 50 | 0
  Cycle 29/Day 1 (Answer to Q1: Yes) | 30.0 |
  Cycle 29/Day 1 (Answer to Q1: No): number analyzed (Participants) | 50 | 0
  Cycle 29/Day 1 (Answer to Q1: No) | 70.0 |
  Cycle 30/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 50 | 0
  Cycle 30/Day 1 (Answer to Q1: Yes) | 32.0 |
  Cycle 30/Day 1 (Answer to Q1: No): number analyzed (Participants) | 50 | 0
  Cycle 30/Day 1 (Answer to Q1: No) | 68.0 |
  Cycle 31/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 49 | 0
  Cycle 31/Day 1 (Answer to Q1: Yes) | 24.5 |
  Cycle 31/Day 1 (Answer to Q1: No): number analyzed (Participants) | 49 | 0
  Cycle 31/Day 1 (Answer to Q1: No) | 75.5 |
  Cycle 32/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 48 | 0
  Cycle 32/Day 1 (Answer to Q1: Yes) | 25.0 |
  Cycle 32/Day 1 (Answer to Q1: No): number analyzed (Participants) | 48 | 0
  Cycle 32/Day 1 (Answer to Q1: No) | 75.0 |
  Cycle 33/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 46 | 0
  Cycle 33/Day 1 (Answer to Q1: Yes) | 28.3 |
  Cycle 33/Day 1 (Answer to Q1: No): number analyzed (Participants) | 46 | 0
  Cycle 33/Day 1 (Answer to Q1: No) | 71.7 |
  Cycle 34/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 44 | 0
  Cycle 34/Day 1 (Answer to Q1: Yes) | 27.3 |
  Cycle 34/Day 1 (Answer to Q1: No): number analyzed (Participants) | 44 | 0
  Cycle 34/Day 1 (Answer to Q1: No) | 72.7 |
  Cycle 35/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 42 | 0
  Cycle 35/Day 1 (Answer to Q1: Yes) | 28.6 |
  Cycle 35/Day 1 (Answer to Q1: No): number analyzed (Participants) | 42 | 0
  Cycle 35/Day 1 (Answer to Q1: No) | 71.4 |
  Cycle 36/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 41 | 0
  Cycle 36/Day 1 (Answer to Q1: Yes) | 26.8 |
  Cycle 36/Day 1 (Answer to Q1: No): number analyzed (Participants) | 41 | 0
  Cycle 36/Day 1 (Answer to Q1: No) | 73.2 |
  Cycle 37/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 37 | 0
  Cycle 37/Day 1 (Answer to Q1: Yes) | 27.0 |
  Cycle 37/Day 1 (Answer to Q1: No): number analyzed (Participants) | 37 | 0
  Cycle 37/Day 1 (Answer to Q1: No) | 73.0 |
  Cycle 38/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 37 | 0
  Cycle 38/Day 1 (Answer to Q1: Yes) | 24.3 |
  Cycle 38/Day 1 (Answer to Q1: No): number analyzed (Participants) | 37 | 0
  Cycle 38/Day 1 (Answer to Q1: No) | 75.7 |
  Cycle 39/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 33 | 0
  Cycle 39/Day 1 (Answer to Q1: Yes) | 30.3 |
  Cycle 39/Day 1 (Answer to Q1: No): number analyzed (Participants) | 33 | 0
  Cycle 39/Day 1 (Answer to Q1: No) | 69.7 |
  Cycle 40/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 32 | 0
  Cycle 40/Day 1 (Answer to Q1: Yes) | 25.0 |
  Cycle 40/Day 1 (Answer to Q1: No): number analyzed (Participants) | 32 | 0
  Cycle 40/Day 1 (Answer to Q1: No) | 75.0 |
  Cycle 41/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 31 | 0
  Cycle 41/Day 1 (Answer to Q1: Yes) | 32.3 |
  Cycle 41/Day 1 (Answer to Q1: No): number analyzed (Participants) | 31 | 0
  Cycle 41/Day 1 (Answer to Q1: No) | 67.7 |
  Cycle 42/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 31 | 0
  Cycle 42/Day 1 (Answer to Q1: Yes) | 25.8 |
  Cycle 42/Day 1 (Answer to Q1: No): number analyzed (Participants) | 31 | 0
  Cycle 42/Day 1 (Answer to Q1: No) | 74.2 |
  Cycle 43/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 29 | 0
  Cycle 43/Day 1 (Answer to Q1: Yes) | 24.1 |
  Cycle 43/Day 1 (Answer to Q1: No): number analyzed (Participants) | 29 | 0
  Cycle 43/Day 1 (Answer to Q1: No) | 75.9 |
  Cycle 44/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 30 | 0
  Cycle 44/Day 1 (Answer to Q1: Yes) | 30.0 |
  Cycle 44/Day 1 (Answer to Q1: No): number analyzed (Participants) | 30 | 0
  Cycle 44/Day 1 (Answer to Q1: No) | 70.0 |
  Cycle 45/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 28 | 0
  Cycle 45/Day 1 (Answer to Q1: Yes) | 25.0 |
  Cycle 45/Day 1 (Answer to Q1: No): number analyzed (Participants) | 28 | 0
  Cycle 45/Day 1 (Answer to Q1: No) | 75.0 |
  Cycle 46/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 29 | 0
  Cycle 46/Day 1 (Answer to Q1: Yes) | 27.6 |
  Cycle 46/Day 1 (Answer to Q1: No): number analyzed (Participants) | 29 | 0
  Cycle 46/Day 1 (Answer to Q1: No) | 72.4 |
  Cycle 47/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 26 | 0
  Cycle 47/Day 1 (Answer to Q1: Yes) | 26.9 |
  Cycle 47/Day 1 (Answer to Q1: No): number analyzed (Participants) | 26 | 0
  Cycle 47/Day 1 (Answer to Q1: No) | 73.1 |
  Cycle 48/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 27 | 0
  Cycle 48/Day 1 (Answer to Q1: Yes) | 29.6 |
  Cycle 48/Day 1 (Answer to Q1: No): number analyzed (Participants) | 27 | 0
  Cycle 48/Day 1 (Answer to Q1: No) | 70.4 |
  Cycle 49/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 24 | 0
  Cycle 49/Day 1 (Answer to Q1: Yes) | 29.2 |
  Cycle 49/Day 1 (Answer to Q1: No): number analyzed (Participants) | 24 | 0
  Cycle 49/Day 1 (Answer to Q1: No) | 70.8 |
  Cycle 50/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 24 | 0
  Cycle 50/Day 1 (Answer to Q1: Yes) | 29.2 |
  Cycle 50/Day 1 (Answer to Q1: No): number analyzed (Participants) | 24 | 0
  Cycle 50/Day 1 (Answer to Q1: No) | 70.8 |
  Cycle 51/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 23 | 0
  Cycle 51/Day 1 (Answer to Q1: Yes) | 26.1 |
  Cycle 51/Day 1 (Answer to Q1: No): number analyzed (Participants) | 23 | 0
  Cycle 51/Day 1 (Answer to Q1: No) | 73.9 |
  Cycle 52/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 103 | 0
  Cycle 52/Day 1 (Answer to Q1: Yes) | 29.2 |
  Cycle 52/Day 1 (Answer to Q1: No): number analyzed (Participants) | 103 | 0
  Cycle 52/Day 1 (Answer to Q1: No) | 70.8 |
  Cycle 53/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 20 | 0
  Cycle 53/Day 1 (Answer to Q1: Yes) | 25.0 |
  Cycle 53/Day 1 (Answer to Q1: No): number analyzed (Participants) | 20 | 0
  Cycle 53/Day 1 (Answer to Q1: No) | 75.0 |
  Cycle 54/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 22 | 0
  Cycle 54/Day 1 (Answer to Q1: Yes) | 36.4 |
  Cycle 54/Day 1 (Answer to Q1: No): number analyzed (Participants) | 22 | 0
  Cycle 54/Day 1 (Answer to Q1: No) | 63.6 |
  Cycle 55/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 17 | 0
  Cycle 55/Day 1 (Answer to Q1: Yes) | 29.4 |
  Cycle 55/Day 1 (Answer to Q1: No): number analyzed (Participants) | 17 | 0
  Cycle 55/Day 1 (Answer to Q1: No) | 70.6 |
  Cycle 56/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 18 | 0
  Cycle 56/Day 1 (Answer to Q1: Yes) | 38.9 |
  Cycle 56/Day 1 (Answer to Q1: No): number analyzed (Participants) | 18 | 0
  Cycle 56/Day 1 (Answer to Q1: No) | 61.1 |
  Cycle 57/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 15 | 0
  Cycle 57/Day 1 (Answer to Q1: Yes) | 20.0 |
  Cycle 57/Day 1 (Answer to Q1: No): number analyzed (Participants) | 15 | 0
  Cycle 57/Day 1 (Answer to Q1: No) | 80.0 |
  Cycle 58/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 103 | 0
  Cycle 58/Day 1 (Answer to Q1: Yes) | 35.3 |
  Cycle 58/Day 1 (Answer to Q1: No): number analyzed (Participants) | 103 | 0
  Cycle 58/Day 1 (Answer to Q1: No) | 64.7 |
  Cycle 59/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 14 | 0
  Cycle 59/Day 1 (Answer to Q1: Yes) | 21.4 |
  Cycle 59/Day 1 (Answer to Q1: No): number analyzed (Participants) | 14 | 0
  Cycle 59/Day 1 (Answer to Q1: No) | 78.6 |
  Cycle 60/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 16 | 0
  Cycle 60/Day 1 (Answer to Q1: Yes) | 37.5 |
  Cycle 60/Day 1 (Answer to Q1: No): number analyzed (Participants) | 16 | 0
  Cycle 60/Day 1 (Answer to Q1: No) | 62.5 |
  Cycle 61/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 13 | 0
  Cycle 61/Day 1 (Answer to Q1: Yes) | 23.1 |
  Cycle 61/Day 1 (Answer to Q1: No): number analyzed (Participants) | 13 | 0
  Cycle 61/Day 1 (Answer to Q1: No) | 76.9 |
  Cycle 62/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 16 | 0
  Cycle 62/Day 1 (Answer to Q1: Yes) | 37.5 |
  Cycle 62/Day 1 (Answer to Q1: No): number analyzed (Participants) | 16 | 0
  Cycle 62/Day 1 (Answer to Q1: No) | 62.5 |
  Cycle 63/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 14 | 0
  Cycle 63/Day 1 (Answer to Q1: Yes) | 21.4 |
  Cycle 63/Day 1 (Answer to Q1: No): number analyzed (Participants) | 14 | 0
  Cycle 63/Day 1 (Answer to Q1: No) | 78.6 |
  Cycle 64/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 14 | 0
  Cycle 64/Day 1 (Answer to Q1: Yes) | 35.7 |
  Cycle 64/Day 1 (Answer to Q1: No): number analyzed (Participants) | 14 | 0
  Cycle 64/Day 1 (Answer to Q1: No) | 64.3 |
  Cycle 65/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 14 | 0
  Cycle 65/Day 1 (Answer to Q1: Yes) | 21.4 |
  Cycle 65/Day 1 (Answer to Q1: No): number analyzed (Participants) | 14 | 0
  Cycle 65/Day 1 (Answer to Q1: No) | 78.6 |
  Cycle 66/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 13 | 0
  Cycle 66/Day 1 (Answer to Q1: Yes) | 30.8 |
  Cycle 66/Day 1 (Answer to Q1: No): number analyzed (Participants) | 13 | 0
  Cycle 66/Day 1 (Answer to Q1: No) | 69.2 |
  Cycle 67/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 12 | 0
  Cycle 67/Day 1 (Answer to Q1: Yes) | 25.0 |
  Cycle 67/Day 1 (Answer to Q1: No): number analyzed (Participants) | 12 | 0
  Cycle 67/Day 1 (Answer to Q1: No) | 75.0 |
  Cycle 68/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 13 | 0
  Cycle 68/Day 1 (Answer to Q1: Yes) | 30.8 |
  Cycle 68/Day 1 (Answer to Q1: No): number analyzed (Participants) | 13 | 0
  Cycle 68/Day 1 (Answer to Q1: No) | 69.2 |
  Cycle 69/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 103 | 0
  Cycle 69/Day 1 (Answer to Q1: Yes) | 25.0 |
  Cycle 69/Day 1 (Answer to Q1: No): number analyzed (Participants) | 103 | 0
  Cycle 69/Day 1 (Answer to Q1: No) | 75.0 |
  Cycle 70/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 13 | 0
  Cycle 70/Day 1 (Answer to Q1: Yes) | 30.8 |
  Cycle 70/Day 1 (Answer to Q1: No): number analyzed (Participants) | 13 | 0
  Cycle 70/Day 1 (Answer to Q1: No) | 69.2 |
  Cycle 71/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 10 | 0
  Cycle 71/Day 1 (Answer to Q1: Yes) | 30.0 |
  Cycle 71/Day 1 (Answer to Q1: No): number analyzed (Participants) | 10 | 0
  Cycle 71/Day 1 (Answer to Q1: No) | 70.0 |
  Cycle 72/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 9 | 0
  Cycle 72/Day 1 (Answer to Q1: Yes) | 22.2 |
  Cycle 72/Day 1 (Answer to Q1: No): number analyzed (Participants) | 9 | 0
  Cycle 72/Day 1 (Answer to Q1: No) | 77.8 |
  Cycle 73/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 9 | 0
  Cycle 73/Day 1 (Answer to Q1: Yes) | 22.2 |
  Cycle 73/Day 1 (No): number analyzed (Participants) | 9 | 0
  Cycle 73/Day 1 (No) | 77.8 |
  Cycle 74/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 8 | 0
  Cycle 74/Day 1 (Answer to Q1: Yes) | 25.0 |
  Cycle 74/Day 1 (Answer to Q1: No): number analyzed (Participants) | 8 | 0
  Cycle 74/Day 1 (Answer to Q1: No) | 75.0 |
  Cycle 75/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 9 | 0
  Cycle 75/Day 1 (Answer to Q1: Yes) | 22.2 |
  Cycle 75/Day 1 (Answer to Q1: No): number analyzed (Participants) | 9 | 0
  Cycle 75/Day 1 (Answer to Q1: No) | 77.8 |
  Cycle 76/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 6 | 0
  Cycle 76/Day 1 (Answer to Q1: Yes) | 16.7 |
  Cycle 76/Day 1 (Answer to Q1: No): number analyzed (Participants) | 6 | 0
  Cycle 76/Day 1 (Answer to Q1: No) | 83.3 |
  Cycle 77/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 8 | 0
  Cycle 77/Day 1 (Answer to Q1: Yes) | 37.5 |
  Cycle 77/Day 1 (Answer to Q1: No): number analyzed (Participants) | 8 | 0
  Cycle 77/Day 1 (Answer to Q1: No) | 62.5 |
  Cycle 78/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 5 | 0
  Cycle 78/Day 1 (Answer to Q1: Yes) | 20.0 |
  Cycle 78/Day 1 (Answer to Q1: No): number analyzed (Participants) | 5 | 0
  Cycle 78/Day 1 (Answer to Q1: No) | 80.0 |
  Cycle 79/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 5 | 0
  Cycle 79/Day 1 (Answer to Q1: Yes) | 20.0 |
  Cycle 79/Day 1 (Answer to Q1: No): number analyzed (Participants) | 5 | 0
  Cycle 79/Day 1 (Answer to Q1: No) | 80.0 |
  Cycle 80/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 4 | 0
  Cycle 80/Day 1 (Answer to Q1: Yes) | 0.0 |
  Cycle 80/Day 1 (Answer to Q1: No): number analyzed (Participants) | 4 | 0
  Cycle 80/Day 1 (Answer to Q1: No) | 100.0 |
  Cycle 81/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 1 | 0
  Cycle 81/Day 1 (Answer to Q1: Yes) | 0.0 |
  Cycle 81/Day 1 (Answer to Q1: No): number analyzed (Participants) | 1 | 0
  Cycle 81/Day 1 (Answer to Q1: No) | 100.0 |
  Cycle 82/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 2 | 0
  Cycle 82/Day 1 (Answer to Q1: Yes) | 0.0 |
  Cycle 82/Day 1 Answer to Q1: (No): number analyzed (Participants) | 2 | 0
  Cycle 82/Day 1 Answer to Q1: (No) | 100.0 |
  Cycle 83/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 1 | 0
  Cycle 83/Day 1 (Answer to Q1: Yes) | 0.0 |
  Cycle 83/Day 1 (Answer to Q1: No): number analyzed (Participants) | 1 | 0
  Cycle 83/Day 1 (Answer to Q1: No) | 100.0 |
  Cycle 84/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 2 | 0
  Cycle 84/Day 1 (Answer to Q1: Yes) | 0.0 |
  Cycle 84/Day 1 (Answer to Q1: No): number analyzed (Participants) | 2 | 0
  Cycle 84/Day 1 (Answer to Q1: No) | 100.0 |
  Cycle 86/Day 1 (Answer to Q1: Yes): number analyzed (Participants) | 1 | 0
  Cycle 86/Day 1 (Answer to Q1: Yes) | 0.0 |
  Cycle 86/Day 1 (Answer to Q1: No): number analyzed (Participants) | 1 | 0
  Cycle 86/Day 1 (Answer to Q1: No) | 100.0 |

18. Secondary Outcome: Agreement Between Central Laboratory ALK FISH and ALK IHC Test Results - Molecular Profiling Evaluable
Description: Agreement between central laboratory anaplastic lymphoma kinase (ALK) fluorescence in situ hybridization (FISH) and ALK immunohistochemistry (IHC) test results is based on analysis of participants in the Molecular Profiling (MP) evaluable population that have an ALK IHC result and an ALK FISH result of either positive or negative only. This MP evaluable population included participants who screen failed, which their ALK test results were negative based on FISH test. Tumor tissue samples from these screen failure participants were consented and kept. These samples served as a part of negative sample set for evaluation of IHC test and/or polymerase chain reaction (PCR) to determine ALK fusion events. Participants with FISH results of uninformative and assay not performed and IHC results of valid IHC status not available were excluded from the analysis of agreement between central laboratory ALK FISH and ALK IHC test results.
Time Frame: During the screening (less than or equal to 28 days prior to dosing)
Population: The MP evaluable population included 812 participants, of which there were 771 participants that had a test result (positive or negative) from both the FISH test and the IHC test.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Positive ALK FISH Status: Participants in the Molecular Profiling Evaluable population that had positive ALK FISH results.
- Participants With Negative ALK FISH Status: Participants in the Molecular Profiling Evaluable population that had negative ALK FISH results.
Arm/Group | Participants With Positive ALK FISH Status | Participants With Negative ALK FISH Status
Number analyzed (Participants) | 238 | 533
Participants
  Participants with Positive ALK IHC Status | 218 [91.4 to 94.9] | 31
  Participants with Negative ALK IHC Status | 20 | 502
Statistical Analysis 1: Comparison: Participants With Positive ALK FISH Status vs Participants With Negative ALK FISH Status; Test type: Superiority or Other; Overall percent agreement = 0.934, 95% CI 2-sided [0.914 to 0.949] — 95% CI for agreement rate is calculated by the Wilson (Score) Confidence Limit method with alpha=0.05
Statistical Analysis 2: Comparison: Participants With Positive ALK FISH Status vs Participants With Negative ALK FISH Status; Test type: Superiority or Other; Kappa = 0.8470, 95% CI 2-sided [0.8065 to 0.8875] — Kappa coefficient is a statistic which measures inter-rater agreement for qualitative (categorical) items

19. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs; All Causalities)
Description: An AE was an untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes: death, initial or prolonged inpatient hospitalization, life-threatening experience, persistent or significant disability/incapacity, congenital anomaly. Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of study medication. Grade 3 and 4 AEs in below table indicated severe AE and life-threatening consequences respectively; Grade 5 indicated death due to AE.
Time Frame: From the first dose of study medication up to 28 days after the last dose of study medication or up to the time that a participant died or received subsequent anticancer treatment (maximum duration between first and last dose: 324.4 weeks)
Population: All randomized participants who received at least 1 dose of study treatment, with treatment assignments designated according to actual study treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 101
Percentage of participants
  AEs | 99.0 | 99.0
  SAEs | 44.2 | 12.9
  Grade 3/4 AEs | 58.7 | 52.5
  Grade 5 AEs | 22.1 | 2.0
  AEs associated with permanent discontinuation | 26.9 | 4.0
  AEs associated with dose reduction | 14.4 | 7.9
  AEs associated with temporary discontinuation | 39.4 | 37.6

20. Secondary Outcome: Percentage of Participants With Treatment-Emergent AEs (Treatment Related)
Description: as for outcome 19
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 104 | 101
Percentage of participants
  AEs | 98.1 | 96.0
  Serious AEs | 8.7 | 3.0
  Grade 3/4 AEs | 43.3 | 40.6
  Grade 5 AEs | 1.9 | 0
  AEs associated with permanent discontinuation | 5.8 | 1.0
  AEs associated with dose reduction | 13.5 | 7.9
  AEs associated with temporary discontinuation | 28.8 | 31.7

ADVERSE EVENTS:
Time Frame: From the first dose of study medication up to 28 days after the last dose of study medication or up to the time that a participant died or received subsequent anticancer treatment (maximum duration between first and last dose: 324.4 weeks).
Description: An event may be categorized as serious in 1 participant and as nonserious in another, or 1 participant may have experienced both serious and nonserious event. Participants who received at least 1 dose of study treatment, with treatment assignments designated according to actual study treatment received during the 1st cycle were analyzed for AEs.
Arm/Group | Crizotinib | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 62/104 | 61/101
Serious Adverse Events (participants affected / at risk) | 46/104 | 13/101
Other Adverse Events (participants affected / at risk) | 103/104 | 100/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib (N=104) | Chemotherapy (N=101)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1
Syncope (Cardiac disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 1
Disease progression (General disorders) | 15 | 1
Impaired healing (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib (N=104) | Chemotherapy (N=101)
Anaemia (Blood and lymphatic system disorders) | 20 | 49
Leukopenia (Blood and lymphatic system disorders) | 12 | 20
Neutropenia (Blood and lymphatic system disorders) | 21 | 37
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 10
Sinus bradycardia (Cardiac disorders) | 13 | 0
Photopsia (Eye disorders) | 7 | 0
Vision blurred (Eye disorders) | 13 | 4
Visual impairment (Eye disorders) | 42 | 8
Abdominal distension (Gastrointestinal disorders) | 11 | 6
Abdominal pain (Gastrointestinal disorders) | 10 | 3
Abdominal pain upper (Gastrointestinal disorders) | 8 | 2
Constipation (Gastrointestinal disorders) | 37 | 27
Diarrhoea (Gastrointestinal disorders) | 63 | 9
Nausea (Gastrointestinal disorders) | 56 | 50
Toothache (Gastrointestinal disorders) | 7 | 0
Vomiting (Gastrointestinal disorders) | 61 | 46
Asthenia (General disorders) | 8 | 10
Chest discomfort (General disorders) | 9 | 4
Chest pain (General disorders) | 16 | 17
Face oedema (General disorders) | 7 | 0
Fatigue (General disorders) | 9 | 17
Oedema (General disorders) | 9 | 1
Oedema peripheral (General disorders) | 27 | 5
Pain (General disorders) | 10 | 6
Pyrexia (General disorders) | 19 | 15
Nasopharyngitis (Infections and infestations) | 22 | 8
Upper respiratory tract infection (Infections and infestations) | 18 | 8
Alanine aminotransferase increased (Investigations) | 69 | 45
Aspartate aminotransferase increased (Investigations) | 62 | 35
Blood albumin decreased (Investigations) | 26 | 16
Blood alkaline phosphatase increased (Investigations) | 10 | 4
Blood bilirubin increased (Investigations) | 5 | 6
Blood creatine phosphokinase increased (Investigations) | 14 | 0
Blood creatinine increased (Investigations) | 9 | 1
Blood lactate dehydrogenase increased (Investigations) | 15 | 1
Gamma-glutamyltransferase increased (Investigations) | 14 | 4
Haemoglobin decreased (Investigations) | 7 | 21
Neutrophil count decreased (Investigations) | 40 | 33
Platelet count decreased (Investigations) | 8 | 27
Protein total decreased (Investigations) | 14 | 3
Red blood cell count decreased (Investigations) | 6 | 9
White blood cell count decreased (Investigations) | 43 | 56
Decreased appetite (Metabolism and nutrition disorders) | 27 | 33
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 16
Hypoproteinaemia (Metabolism and nutrition disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 6
Dizziness (Nervous system disorders) | 28 | 11
Taste disorder (Nervous system disorders) | 6 | 0
Headache (Nervous system disorders) | 29 | 9
Hypoaesthesia (Nervous system disorders) | 9 | 2
Paraesthesia (Nervous system disorders) | 7 | 4
Insomnia (Psychiatric disorders) | 14 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 8
Rash (Skin and subcutaneous tissue disorders) | 12 | 7
Phlebitis (Vascular disorders) | 1 | 8
Bradycardia (Cardiac disorders) | 6 | 0
Pneumonia (Infections and infestations) | 6 | 0
Blood creatine phosphokinase MB increased (Investigations) | 6 | 0
Lymphocyte count decreased (Investigations) | 8 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 0
Hypertension (Vascular disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.